CLINICAL TRIAL: NCT02264041
Title: The Effect of Cytochrome P 450 3A4 Inhibition by Itraconazole on the Single Oral Dose Pharmacokinetics of Cilobradine (an Open-label, Randomised, Single-dose, Two-way Crossover Study)
Brief Title: Effect of Cytochrome P 450 3A4 Inhibition by Itraconazole on the Single Oral Dose Pharmacokinetics of Cilobradine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 503.213
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — cilobradine; Itraconazole

ARMS (4):
- Cilobradine, low dose plus itraconazole (Experimental): Pre-study
  Interventions: Drug: Cilobradine, low dose; Drug: Itraconazole
- Cilobradine, low dose (Active Comparator): Pre-study
  Interventions: Drug: Cilobradine, low dose
- Cilobradine, high dose plus itraconazole (Experimental): main study
  Interventions: Drug: Cilobradine, high dose; Drug: Itraconazole
- Cilobradine, high dose (Active Comparator): main study
  Interventions: Drug: Cilobradine, high dose

INTERVENTIONS:
Drug: Cilobradine, low dose
  Arms: Cilobradine, low dose; Cilobradine, low dose plus itraconazole
Drug: Cilobradine, high dose
  Arms: Cilobradine, high dose; Cilobradine, high dose plus itraconazole
Drug: Itraconazole
  Other Names: Sempera®
  Arms: Cilobradine, high dose plus itraconazole; Cilobradine, low dose plus itraconazole

SUMMARY:
Study to investigate the effect of cytochrome P 450 3A4 inhibition by itraconazole on the single dose pharmacokinetics of cilobradine

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests

   1.1 No finding deviating from normal and of clinical relevance

   1.2 No evidence of a clinically relevant concomitant disease
2. Age ≥21 and Age ≤55 years
3. BMI ≥18.5 and BMI < 30 kg/m2 (Body Mass Index)
4. Resting pulse rate (PR; after 10 min. in the supine position) of more than 55 bpm
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, ophthalmological, or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. History of relevant orthostatic hypotension, fainting spells or blackouts.
4. Chronic or relevant acute infections
5. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
6. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
7. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial.
8. Participation in another trial with an investigational drug within two months prior to administration or during the trial
9. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
10. Inability to refrain from smoking on trial days
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2004-01; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 56 hours after administration of Cilobradine
Maximum measured concentration of the analyte in plasma (Cmax) | up to 56 hours after administration of Cilobradine

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | up to 56 hours after administration of Cilobradine
Time from dosing to Cmax (Tmax) | up to 56 hours after administration of Cilobradine
Terminal rate constant in plasma (λz) | up to 56 hours after administration of Cilobradine
Terminal half-life of the analyte in plasma (t1/2) | up to 56 hours after administration of Cilobradine
Mean residence time of the analyte in the body after p.o. administration (MRTpo) | up to 56 hours after administration of Cilobradine
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | up to 56 hours after administration of Cilobradine
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | up to 56 hours after administration of Cilobradine
Amount of parent compound excreted in urine with zero to 72 h in % of dose (fe0-tz) | up to 72 hours after administration of Cilobradine
Renal clearance of cilobradine (CLR,0-tz) | up to 72 hours after administration of Cilobradine
Number of subjects with adverse events | up to 46 days
Occurrence of visual phenomena | up to 46 days
  questionnaire
Number of subjects with clinically relevant findings in vital signs | up to 32 days
  blood pressure, pulse rate
Number of subjects with clinically relevant findings in laboratory tests | up to 32 days
Number of subjects with clinically relevant findings in 12-lead electrocardiogram | up to 32 days
Assessment of tolerability by investigator on a 4-point scale | within 8 days after last PK sampling